CLINICAL TRIAL: NCT02246868
Title: An Open Study to Investigate the Safety and Efficacy of Optivate® in Severe Haemophilia A Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 8VWFSE
Record Dates: First submitted 2014-09-02; First posted 2014-09-23 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — optivate; Factor VIII

ARMS (1):
- Optivate® (Experimental): Optivate® (Human Coagulation Factor VIII)
  Interventions: Biological: Optivate® (Human Coagulation Factor VIII)

INTERVENTIONS:
Biological: Optivate® (Human Coagulation Factor VIII)

SUMMARY:
The main objectives of this study are to compare the first and second recovery assessments and recovery when a subject changed batch and to assess whether haemostasis was achieved with Optivate® when treating a bleed. The secondary objectives are to evaluate the clinical tolerance and safety of Optivate®.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent with severe Haemophilia A without inhibitor to FVIII, at least 12 years of age, currently receiving FVIII concentrates and have more than 150 exposures. Subjects who require elective surgergy within 6 months of starting on OPTIVATE® are permitted to be included in this study providing that the surgery could be performed using OPTIVATE® as FVIII cover.

Exclusion Criteria:

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Incremental Recovery | Comparison of Baseline with 3 months post-baseline

CONTACTS AND LOCATIONS:
Locations (11):
- Poland (6):
  - Klinika Haematologii, Akademia Medyczna w Bialymstokiu, ul., Bialystok
  - Klinika Haematologii, Akademia Medyczna w Gdansku, u., Gdansk
  - Klinika Haematologii, Akademia Medyczna w Lodzi, ul., Lodz
  - Klinika Haematologii, Akademia Medyczna w Lublinie, ul., Lublin
  - Klinika Haematologii, Akademia Medyczna w Poznaniu, ul., Poznan
  - Klinika Haematologii, Akademia Medyczna w Wroclawiu, ul., Wroclaw
- United Kingdom (5):
  - Haemophilia Centre, Addenbrooke's Hospital, Hills Road, Cambridge
  - Haemophilia Centre, University Department of Haemophilia Manchester Royal Infirmary, Manchester
  - Haemophilia Centre, University Hospital, Queen's Medical Centre, Clifton Boulevard, Nottingham
  - Sheffield Haemophilia & Thrombosis Centre, Royal Hallamshire Hospital, Glossop Road, Sheffield
  - Haemophilia Centre, Southampton General Hospital, Tremona Road, Southampton

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk